CLINICAL TRIAL: NCT03688841
Title: Bridged Vacuum Assisted Closure (VAC) With Compression vs. Compression Therapy in the Management of Venous Leg Ulcers: A Prospective Randomised Controlled Trial
Brief Title: Negative Pressure Vs. Compression in Venous Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Vascular Institute, Ireland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BVACC-CCD
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Varicose Ulcer
Keywords: Varicose ulcer; Compression Therapy; Negative Pressure; Vacuum Assisted Closure
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: This is a randomised, parallel group, active-control trial, with patients randomised in a 1:1 ratio to one of two treatment arms.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the obvious differences between the intervention and comparator, it is impossible to blind the participants or the care providers.
  However, the investigator, the outcomes assessor and statistician are blinded to treatment received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bridged V.A.C.® with compression therapy (Experimental): A vacuum assisted closure device will be placed on the ulcer. A compression dressing will be placed over the V.A.C.® device
  Interventions: Device: Bridged V.A.C.® with compression therapy
- Conventional compression therapy (Active Comparator): A Coban™ Lite compression dressings with underlying non-adherent wound contact layer (WCL) dressings will be applied and changed once to three times per week (dependant on exudate).
  Interventions: Device: Conventional Compression Therapy

INTERVENTIONS:
Device: Bridged V.A.C.® with compression therapy — Patients randomised to receive Bridge VAC with compression dressings will be managed using ActiV.A.C. Therapy unit, with a continuous pressure of 125mmHg. A V.A.C.® Granufoam™ Bridge Dressing will be used instead of the tube connector. A Coban™ Lite compression dressing will be placed over the VAC dressing. The Bridge connector of the VAC will be used to tunnel underneath the Coban™ Lite till the upper edge of the dressing.
  Arms: Bridged V.A.C.® with compression therapy
Device: Conventional Compression Therapy — Patients randomised to receive compression dressings will be managed using Coban™ Lite compression dressings with underlying non-adherent wound contact layer (WCL) dressings. Under the supervision of the investigating clinician, the dressings will be applied by a wound care specialist nurse and changed once to three times per week (depending on amount of exudate), until full ulcer healing or up to 12 weeks.
  Arms: Conventional compression therapy

SUMMARY:
This study randomises patients with venous leg ulcers, to be managed either using conventional compression bandages or a bridged vacuum assisted closure system under compression.

DETAILED DESCRIPTION:
Venous ulcers are characterised by a cyclical pattern of healing and recurrence, with recurrence rates between 45 and 70% at one year. Venous leg ulceration has been identified as a common source of morbidity and reduced quality of life, especially in the elderly population. Non-healing ulcers place the patient at a much higher risk for lower extremity amputation.

Compression therapy is currently recognised as the main treatment for venous leg ulcers. External compression is applied as a therapy for venous leg ulcers, in an attempt to reverse the increased hydrostatic pressure in the veins.

The application of negative pressure to successfully treat and aid in the healing of open wounds has been studied extensively for decades, demonstrating favourable clinical results. However, there is a lack of evidence in the literature regarding the use of VAC in venous ulcers.

The combination of negative pressure therapy and compression therapy is theorized to provide the benefits of both individual therapies. As such, the utilization of the Bridge VAC under a compression dressing is expected to expedite the healing of venous ulcers.

The investigators aim to randomise patients with venous ulcers to either be managed using conventional compression dressings or combined bridge vacuum assisted closure with compression dressings.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more
* Provide written informed consent
* Venous ulcer present, greater than 10cm2 in surface area
* A C6 grading in the CEAP classification

Exclusion Criteria:

Pregnant (confirmed by β-HCG analysis). Female patients of childbearing potential are advised to adhere to an appropriate form of contraception, and those unwilling to follow contraceptive advice are excluded from the study

* Involvement in another clinical trial in the previous six months
* Legal incapacity
* Patient is bed-ridden or immobile
* Ulcer smaller than 10cm2 in surface area
* Ischaemic ulcer/s present
* Diabetic ulcer/s present
* Malignant ulceration/s present
* Ulcer exposing bone or tendon
* Osteomyelitis
* Pseudomonas infection
* Presence of gangrene
* Deep venous thrombosis (DVT) present
* Connective tissue disease present
* Presence of any illness that could limit long-term compliance (e.g. epilepsy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Time to healing | 12 weeks
  The time taken for complete closure of the index ulcer or till the wound is judged suitable for skin grafting

SECONDARY OUTCOMES:
Proportion of ulcers healed | 12 weeks
  The proportion of index ulcers fully healed
Ulcer recurrence | 12 months
  Wound recurrence rates at six weeks, and three, six and 12 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Sultan, MD, Principal Investigator — Western Vascular Institute, Ireland; Wael Tawfick, MD, Principal Investigator — Western Vascular Institute, Ireland
Locations (1):
- Department of Vascular Surgery, Western Vascular Institute, Galway University Hospital, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No
IPD of primary and secondary outcomes, could be made available to other researchers by request, while maintaining participant confidentiality